CLINICAL TRIAL: NCT04234685
Title: Determining the Effectiveness of a Novel Phototherapy for the Treatment of Knee Osteoarthritis: a Pilot Randomized Controlled Trial
Brief Title: Determining the Effectiveness of a New Phototherapy Treatment for the Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan Miller, PT, PhD (Other)
Collaborators: Invitalize (Unknown)
Responsible Party: Sponsor-Investigator, Jordan Miller, PT, PhD, Associate Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REH-708-17
Record Dates: First submitted 2019-03-28; First posted 2020-01-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Educational Status; Self-Management; Exercise; Resistance Training; Circuit-Based Exercise

STUDY DESIGN:
Intervention Model Description: Double (patient and investigator) blind, parallel group, pilot randomized control trial with 1:1 allocation ratio to HIPL Therapy™ or placebo control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized using a computer generated random number generator. The allocation sequence will be recorded on cards placed in sealed, opaque envelopes. Allocation will be concealed until after the initial assessment is completed. At this point the research assistant (physiotherapist) will open the sealed envelope, which will indicate either Group A or Group B, then initiate the phototherapy session by pressing on the corresponding button for Group A or B, which will deliver the appropriate phototherapy intensity for the respective group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIPL Therapy™ group (Experimental): All participants from both groups will take part in a standardized education and exercise intervention as suggested by best evidence. These sessions will be 20-30 minutes in length and will take place twice weekly for four weeks (8 sessions).
  The HIPL Therapy™ group will receive phototherapy in addition to the education and exercise intervention twice weekly for four weeks. Participants will lay in a relaxed position on a therapy plinth with the light applied using the Invitalizer 2.0. The phototherapy will illuminate the affected knee for 20 minutes. In the case of bilateral knee OA, the treatment time will be doubled and applied to both knees. The knee will be positioned at a determined distance from the lamp with an intensity setting of 150 mW/cm2.
  Interventions: Device: High Intensity Physio Light Therapy (HIPL Therapy™); Behavioral: Education; Behavioral: Aerobic Exercise; Behavioral: Resistance Exercise
- Placebo Control group (Placebo Comparator): All participants from both groups will take part in a standardized education and exercise intervention as suggested by best evidence. These sessions will be 20-30 minutes in length and will take place twice weekly for four weeks (8 sessions).
  The placebo control group will also receive phototherapy in addition to the education and exercise intervention twice weekly for four weeks, in the same setting as the HIPL Therapy™ group and for the same duration. However, the intensity setting will be set at 5 mW/cm2, a dosage, at which there is no therapeutic benefit expected, but the light will still be visible to the participant.
  Interventions: Behavioral: Education; Behavioral: Aerobic Exercise; Behavioral: Resistance Exercise; Device: Placebo Physio Light Therapy (HIPL Therapy™)

INTERVENTIONS:
Device: High Intensity Physio Light Therapy (HIPL Therapy™) — HIPL Therapy™ is an advanced phototherapy method that utilizes an emission wavelength spectrum that has been optimized for treatment of musculoskeletal disorders (MSD) such as OA.
  Other Names: Invitalizer 2.0 (Invitalize, Kitchener Ontario)
  Arms: HIPL Therapy™ group
Behavioral: Education — Participants will take part in education on osteoarthritis, pain neurophysiology, and self-management strategies with the treating physiotherapist. The education will take place during the lab visits and will be brief (5-10 minutes at each session).
  Other Names: Self-management, pain neurophysiology
Behavioral: Aerobic Exercise — Participants will develop an individualized walking program. The goal will be to walk 30 minutes 5 times/week if able. For all participants who are unable to achieve this walking, they will be provided with a progressive walking program that starts at their baseline (the distance they can walk without being sore an hour later; and without feeling like they will be unable to perform their usual activities of daily living because of the walk). They will be encouraged to then progress by 10-20% each week. Participants will be asked to use a provided walking log to keep track of their progress.
  Other Names: Walking program
Behavioral: Resistance Exercise — Participants will also be instructed how to perform a series of six exercises: squat, step-up, lunge, single leg stance, knee flexion/extension, and resisted hamstring curl. The exercise technique and dosage will be tailored to the individual's current abilities. For example, if someone is unable to squat down to the level of a chair and return to standing, the chair height will be raised until the participant is able to perform the activity. The participants will begin by being asked to complete one set of 8-12 repetitions of each exercise, once daily, then progress to two or three sets daily as able. They will perform the exercises twice/week in the lab where they will receive support for problem solving and progression. Participants will be asked to use a provided exercise log to keep track of their progress.
  Other Names: Strength training, circuit training
Device: Placebo Physio Light Therapy (HIPL Therapy™) — Phototherapy delivered at an intensity of 5 mW/cm2, a dosage at which there is no therapeutic benefit expected, but the light will still be visible to the participant.
  Other Names: Control
  Arms: Placebo Control group

SUMMARY:
Light therapy (phototherapy) has previously been shown to help reduce pain for people with musculoskeletal pain conditions, such as knee osteoarthritis (OA). A new phototherapy has been developed that allows for customizing the intensity of light based on patient characteristics, such as the patient size and skin type. This new phototherapy approach needs to be evaluated to determine its effects. This study has been planned to determine how effective the new phototherapy is, but first it needs to be determined whether the study plans are feasible. This study will determine the feasibility of the full study by pilot testing the methods for the full trial with a group of 20 people with knee osteoarthritis. Participants will be randomly assigned to either receive the new phototherapy approach or a placebo phototherapy twice/week for four weeks. Pain and function will be measured over the four week treatment period and 12-weeks follow-up.

DETAILED DESCRIPTION:
Invitalize has developed the High Intensity Physio Light (HIPL) Therapy™, a phototherapy method that utilizes an emission wavelength spectrum that has been identified for treatment of musculoskeletal disorders (MSD) such as OA.

Design: Double (patient and investigator) blind, parallel group, pilot randomized control trial with 1:1 allocation ratio to HIPL Therapy™ or placebo control.

Recruitment: For the pilot, 20 adults who have been diagnosed with knee osteoarthritis (OA) of any duration will be recruited to participate in this study at Queen's University. Participants will be recruited from two primary care practices in Kingston, Ontario.

Randomization and allocation concealment: Participants will be randomized to either the placebo or control group using a computer generated random number generator. The allocation sequence will be recorded on cards placed in sealed, opaque envelopes. Allocation will be concealed until after the initial assessment is completed. Patients and investigators will remain blinded throughout the trial.

The HIPL Therapy™ group will receive phototherapy in addition to an education and exercise intervention with a physiotherapist twice weekly for four weeks. Participants will lay in a relaxed position on a therapy plinth with the light applied to the affected knee for 20 minutes. In the case of bilateral knee OA, the treatment time will be doubled and applied to both knees with an intensity setting aimed at delivering 150 mW/cm2.

The control group will receive the same education and exercise intervention, as well as 20 minutes of phototherapy twice weekly for four weeks. However, the intensity setting will be set at 5 mW/cm2, a dosage at which there is no therapeutic benefit expected, but the light will still be visible to the participant.

All participants will complete brief questionnaires at each visit and will complete functional assessments and pressure point testing at the initial, fourth and final visits. Participants will complete online questionnaires at the 8-, 12- and 16-week time points as well.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults (>18 years of age)
* Provided with a diagnosis of knee OA by a physician
* Self-report of having experienced pain and disability related to knee OA for at least 6 months.

Exclusion Criteria:

* Skin conditions in which application of phototherapy may be contra-indicated (skin cancer, people receiving radiation therapy)
* History of total joint arthroplasty of the affected knee
* Red flags suggestive of non-musculoskeletal etiology (i.e. fever/chills, unrelenting night pain, multi-segmental or bilateral loss of sensation, sudden unexplained weight loss).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Baseline
  The feasibility of patient recruitment will be determined by the overall recruitment rate. The full trial will be considered feasible with our current recruitment methods if, during the pilot study, an average recruitment rate of at least 3 patients per week is achieved. This recruitment rate will allow us to exceed the 168 participants needed for a fully powered trial in a 56 week recruitment period. The findings of this study will inform whether this preliminary plan is feasible or if additional sites are needed.
Feasibility of Assessment Procedures: completion rate | Through study completion (16 weeks)
  Feasibility of the assessment procedures will be measured by completion rate of outcome measures. As recommended for pilot studies, we set criteria a priori for acceptable completeness and considered >80% of all assessment items completed.
Retention Rate | Through study completion (16 weeks)
  Retention will be assessed by attrition rate, with <20% attrition at 3-month follow-up (16 weeks) considered indicative of feasibility with our current protocol.
Feasibility of Research Assistant (RA) Training: rating | Baseline
  Feasibility of training the RA who will implement the phototherapy intervention will be evaluated a rating of self-efficacy (0-10) for delivering the intervention, where a lower score would indicate a lower rating of preparedness for delivering the intervention and a higher score would indicate a higher rating of preparedness to deliver the intervention.
Monitoring Treatment Fidelity | Through study completion (16 weeks)
  Fidelity was measured through an audit of the fidelity checklist and reported as a proportion of intervention components delivered in alignment with the protocol. An a-priori acceptable level of fidelity was considered 80% for each component of the intervention among participants that attend each visit.

SECONDARY OUTCOMES:
Change in Sensitivity to Physical Activity (SPA) | Baseline, 2 weeks, 4 weeks (1st, 4th and 8th clinic visits)
  Change in SPA will be measured using the change in reported knee pain throughout the 6MWT. Pain intensity will be measured each minute throughout the 6MWT using a 100mm visual analogue scale (VAS) with anchors including no pain (0) to worst imaginable pain (100mm). The SPA index will be the difference between the peak pain intensity during the 6MWT and the baseline pain intensity at rest.
  Pain during physical activity will be the primary outcome measure for the full trial, measured using the change in SPA.
Change in Physical Function | Baseline, 2 weeks, 4 weeks (1st, 4th and 8th clinic visits)
  Change in physical function will be measured using the 6-minute walk test (6MWT). The 6MWT is a test of walking speed/aerobic capacity/endurance. It involves walking continuously on a 30-meter walkway for 6 minutes. The score on the test is the distance walked.
Change in Pain Intensity: VAS | Each clinical visit (twice per week for four weeks)
  Change in pain intensity will be measured using a 100mm visual analogue scale (VAS) with anchors including no pain (0) to worst imaginable pain (100mm). Participants will be asked to report their pain intensity at its worst in the past 24 hours, at its best in the past 24 hours, their average pain and their pain right now.
Change in Self-Reported Function | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Change in self-reported function - physical function will be measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) physical function subscale (0 to 68) with higher scores indicating greater functional limitations. The WOMAC physical function subscale uses a series of questions about functional tasks answered on a four-point Likert scale.
Monitoring Exercise Adherence | Through study completion (16 weeks)
  Adherence to prescribed exercise will be measured using a self-report diary of all exercises prescribed.
Global Rating of Change in Pain | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Global rating of change in pain will be measured using an 11-point global rating of change (GROC) scale (-5 to +5, where -5 is much worse and +5 is much better), as has been recommended in the literature for self-reported rating of change
Global Rating of Change in Functional Abilities | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Global rating of change in functional abilities will be measured using an 11-point global rating of change (GROC) scale (-5 to +5, where -5 is much worse and +5 is much better), as has been recommended in the literature for self-reported rating of change
Global Rating of Change in Satisfaction with Care | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Global rating of change in satisfaction with care will be measured using an 11-point global rating of change (GROC) scale (-5 to +5, where -5 is very dissatisfied and +5 is very satisfied), as has been recommended in the literature for self-reported rating of change
Change in Pressure Pain Threshold: Newtons (N) | Baseline and 4 weeks (1st and 8th clinic visits)
  Change in pressure pain threshold will be assessed as follows: pressure will be applied at nine predetermined points around the knee using a handheld pressure algometer. Participants will be asked to report the moment the pressure switches from comfortable pressure to slightly unpleasant pain. The pressure pain threshold will be recorded in Newtons (N). This is measured as a process outcome to determine if it relates to SPA.
Adverse Events | 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Adverse events will be recorded using an adverse events questionnaire that is reported consistently with reporting guidelines and asks: 1) if the patient has experienced any events as a result of any of the treatments received (yes/no); 2) how long the event lasted (hours or days); 3) How severe the adverse event was (0-10 scale); 4) what adverse events were experienced. Any serious adverse events will be addressed immediately by referral to the most appropriate member of the primary health care team.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vader K, Abebe AB, Chala MB, Varette K, Miller J. Determining the feasibility of a trial to evaluate the effectiveness of phototherapy versus placebo at reducing pain during physical activity for people with knee osteoarthritis: a pilot randomized controlled trial. Pilot Feasibility Stud. 2020 Nov 26;6(1):186. doi: 10.1186/s40814-020-00729-4. PMID 33292671